CLINICAL TRIAL: NCT07029906
Title: pErsonalised Nocebo Assessment of Beta-blockEr Symptoms in Heart Failure
Acronym: ENABLE-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: PG/22/10715
Record Dates: First submitted 2025-04-29; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Side-Effect; Heart Failure
Keywords: Side-effect; Beta-blocker; Nocebo; Heart Failure Reduced Ejection Fraction; HFrEF; Heart Failure
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic | interventions — Bisoprolol

STUDY DESIGN:
Intervention Model Description: Prospective, N-of-1 study of symptoms in 150 participants with heart failure with reduced ejection fraction. Each participant will follow an individualised protocol after randomly being assigned to a regime.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Blinded bisoprolol tablets (Experimental): The protocol includes a randomised, blinded nine week phase in which participants take either bisoprolol, no tablets or placebo. They will be randomly assigned to take three weeks in total of blinded bisoprolol tablets.
  Interventions: Drug: Bisoprolol 2.5 mg
- Blinded placebo (Placebo Comparator): Participants will be randomly assigned to take three weeks of blinded placebo tablets. They will be unaware as to whether they are consuming bisoprolol or placebo in this phase.
  Interventions: Drug: Placebo
- No tablet (No Intervention): There will be three weeks in total during the randomised phase in which patients do not consume any tablets.

INTERVENTIONS:
Drug: Bisoprolol 2.5 mg — Active bisoprolol 2.5mg tablets
  Arms: Blinded bisoprolol tablets
Drug: Placebo — Blinded placebo for a total of 3 weeks
  Arms: Blinded placebo

SUMMARY:
Beta-blocker tablets are an effective treatment for heart failure that make people live longer and reduce the need to be admitted to hospital. Many patients who are at high risk of death are prescribed beta-blockers, but later choose to stop taking them because of symptoms that they perceive to be side-effects. Some patients' symptoms may genuinely be side-effects due to the beta-blocker tablets, but, in reality, many of the symptoms which may lead to people stopping beta-blockers are actually experienced at similar rates compared to placebo. The symptoms may be caused by heart failure itself, or the expectation that they will have a side effect when they take a tablet (the nocebo effect). There is a need to be able to identify the majority of patients who aren't actually having side-effects so that they can restart beta-blockers and not miss out on life-prolonging treatment. To answer this question reliably and with high precision requires a personalised approach with an 'N-of-1' study. This study will measure participants' symptoms in three scenarios: taking a beta-blocker tablet (bisoprolol 2.5mg) or a placebo tablet or no study medication in a randomised order.

The primary aim of this study is to determine, for an individual, whether the adverse effects of beta-blockade in heart failure are genuine. Specifically, the objectives are:

1. To determine the proportion of a patient's symptoms that are due to taking beta-blocker tablets, and the proportion that are due to the expectation that the treatment will cause symptoms (the nocebo effect).
2. To determine whether, on average, symptoms are worse when taking beta-blocker compared to placebo tablets or no treatment.
3. To determine whether on average symptom intensity associated with beta-blockade decreases after receiving a report on how much of their symptoms are due to the beta-blocker.

Throughout the protocol participants report daily the intensity of the symptom that previously led to their beta-blocker cessation via a smartphone app. Participants will report weekly their adherence, general heart failure symptoms and quality of life. In this way the investigators will discover, for an individual patient, the proportion of their symptom that is due to the beta-blocker tablet, and whether knowing their personalised results helps them to restart beta-blocker tablets.

DETAILED DESCRIPTION:
Method:

ENABLE-HF is a prospective, N-of-1 randomised study of symptoms in participants with HFrEF. The study population will be patients who have an indication for oral beta-blockade due to HFrEF, and are currently not taking any beta-blockers licenced for HFrEF, having previously tried and stopped taking them due to perceived symptoms that they and/or their clinician(s) attributed to the beta-blocker(s).

Participants' suitability will be assessed by a detailed clinical history, clinical examination and review of their medical history to confirm the diagnosis of HFrEF, indication for beta-blocker therapy and that they are currently not taking it. The inclusion and exclusion criteria will be applied. At enrolment, a researcher will generate and allocate an unused randomisation code to the participant. This will also determine the contents of their 9 study bottles to be taken in Phase 2. The participant will then be provided with packs containing all phases' medications, and a smartphone if required.

The study protocol has three main phases:

(i) Phase 1 - a two week, open-label period of 2.5mg bisoprolol daily

(ii) Phase 2 - a nine week double blinded n-of-1 phase consisting of three separate weeks of daily bisoprolol 2.5mg, three separate weeks of daily matched placebo, and three separate weeks of no study tablet. The order of the nine weeks will be randomised at the outset.

(iii) Phase 3 - another two week, open-label period of 2.5mg bisoprolol daily.

Patients will report the intensity of the main symptom that led to them stopping beta-blocker tablets using a smartphone app daily. They will answer a weekly quality-of-life questionnaire. In this way the investigators will discover, for an individual patient, the proportion of their symptom that is due to the beta-blocker tablet, and whether knowing their personalised results helps them to restart beta-blocker tablets.

Each participant will receive a personalised report of their symptom scores from the n-of-1 Phase 2 period. At this point patients and researchers will be unblinded and patients will be counselled by a Cardiologist from research team about what these results mean and how much of their perceived side-effects are attributable to the beta-blocker. These findings will be delivered using pre-determined standardised language.

This study will develop a novel method to provide patients with HFrEF who are currently missing out on the prognostic benefits of beta-blockers with personalised information about their symptom aetiology. It is expected that getting these personalised results will improve long-term beta-blocker adherence in heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with index LVEF <40%
* Not currently taking beta-blocker tablets
* Previously tried one of beta-blocker tablet, and stopped taking it due to symptoms attributed to the beta-blocker
* Consenting to participate in the study

Exclusion Criteria:

* Documented anaphylaxis to beta-blockers
* Clinical contraindication to Bisoprolol including (but not limited to):

  1. Asthma requiring BTS treatment step 3 or higher
  2. Marked bradycardia (<50 bpm)
  3. Symptomatic hypotension (systolic BP <85mmHg)
  4. Metabolic acidosis
  5. Phaeochromocytoma
  6. 1st degree heart block with PR interval >250ms
  7. 2nd degree or complete heart block
  8. Sick sinus syndrome
  9. Acute pulmonary oedema
* Life expectancy <1 year
* Patient refusal or inability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Nocebo Fraction | From start of protocol to end of second open-label beta-blocker phase, an average of 15 weeks
  For each participant, we will primarily calculate the 'nocebo fraction'. This is a measure of the proportion of an individual patient's symptoms which are due to beta-blocker and which are due to the nocebo effect. It is calculated by measuring and averaging the daily symptom intensity (scored from 0 to 100) when taking:
  [A] beta-blocker tablet
  [B] placebo (blank) tablet
  [C] no tablet

SECONDARY OUTCOMES:
Difference in Symptom Intensity Scores Between Beta-Blocker and Placebo | From start of protocol to end of second open-label beta-blocker phase, an average of 15 weeks
  At enrolment, patients will establish one primary symptom that previously resulted in their cessation of taking beta-blockade. This intensity of this symptom will be enquired about on a daily basis through all phases of the trial. To establish how beta-blockers impact this symptom intensity, the difference in average symptom intensity (scored from 0-100) taking a beta-blocker will be compared to that whilst taking a placebo across the population. Symptom intensity will be measured using the self-reported symptom scores that participants report in the app.
Change in Symptom Intensity Scores after Receiving n-of-1 Personalised Results | From start of protocol to end of second open-label beta-blocker phase, an average of 15 weeks
  To determine whether average symptom scores are affected by insights from the n-of-1 period, we will compare the average symptom scores during open-label beta-blocker treatment before the n-of-1 period to those after the n-of-1 period, following receipt of a personalised symptom report. Statistical significance will be assessed using a comparison of means, such as Student's t-test, or non-parametric alternatives if the data are not normally distributed.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Cole, MB BChir, Principal Investigator — Imperial College NHS Trust
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barron AJ, Zaman N, Cole GD, Wensel R, Okonko DO, Francis DP. Systematic review of genuine versus spurious side-effects of beta-blockers in heart failure using placebo control: recommendations for patient information. Int J Cardiol. 2013 Oct 9;168(4):3572-9. doi: 10.1016/j.ijcard.2013.05.068. Epub 2013 Jun 21. PMID 23796325
- [Background] Cole GD, Patel SJ, Zaman N, Barron AJ, Raphael CE, Mayet J, Francis DP. "Triple therapy" of heart failure with angiotensin-converting enzyme inhibitor, beta-blocker, and aldosterone antagonist may triple survival time: shouldn't we tell patients? JACC Heart Fail. 2014 Oct;2(5):545-8. doi: 10.1016/j.jchf.2014.04.012. PMID 25301161
- [Background] Zaman S, Zaman SS, Scholtes T, Shun-Shin MJ, Plymen CM, Francis DP, Cole GD. The mortality risk of deferring optimal medical therapy in heart failure: a systematic comparison against norms for surgical consent and patient information leaflets. Eur J Heart Fail. 2017 Nov;19(11):1401-1409. doi: 10.1002/ejhf.838. Epub 2017 Jun 8. PMID 28597606
- See also: ENABLE-HF Website — https://www.enablehf.net/home